CLINICAL TRIAL: NCT01608165
Title: CONSERVE: a Feasibility Study for a Multicentre Randomised Controlled Trial to Compare Surgery (Partial Nephrectomy) With Needle Ablation Techniques (Radiofrequency Ablation/Cryotherapy) for the Treatment of People With Small Renal Masses (4cm)
Brief Title: A Feasibility Study for a Multicentre Randomised Controlled Trial to Compare Surgery With Needle Ablation Techniques in People With Small Renal Masses (4cm)
Acronym: CONSERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CRUK/11/036; CRUK/11/036 (Other Grant/Funding Number: Cancer research UK); ISRCTN23852951 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Renal Cancer
Keywords: Small renal cancer mass
MeSH Terms: conditions — Kidney Neoplasms | interventions — Surgical Procedures, Operative; Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Partial nephrectomy (Other): Patients randomised to this arm will undergo a partial nephrectomy
  Interventions: Procedure: Surgical treatment for renal mass
- Radiofrequency ablation (Other): Patients randomised to this arm will undergo radiofrequency ablation
  Interventions: Procedure: Percutaneous Radiofrequency ablation
- cryoablation (Other): Patients randomised to this arm will undergo cryoablation
  Interventions: Procedure: Laparascopic or percutaneous cryoablation

INTERVENTIONS:
Procedure: Surgical treatment for renal mass — Patients will be randomised to receive a partial nephrectomy as treatment for their renal cancer mass
  Arms: Partial nephrectomy
Procedure: Percutaneous Radiofrequency ablation — Patients may be randomised to undergo a radiofrequency ablation treatment for their renal cancer mass
  Arms: Radiofrequency ablation
Procedure: Laparascopic or percutaneous cryoablation — Patients may be randomised to undergo cryoablation as treatment for their renal cancer mass
  Arms: cryoablation

SUMMARY:
The number of people diagnosed with kidney cancer has doubled over the past 20 years, making it the eight most common cancer in the UK. Most tumours are less than 4cm in size, but over 80% of these are malignant (cancerous) and if left untreated, will slowly grow and spread. Current standard treatment for these small kidney cancers is to remove the diseased part of the kidney in an operation called a partial nephrectomy, but this can be quite a difficult operation. Because of the small tumour size and difficulties with the operation, other treatments have been developed to destroy the tumours. These treatments include radiofrequency ablation, which means that the tumour is destroyed by heat, and cryoablation, which means that the tumour is frozen and destroyed.

Although removing the part of the diseased kidney in an operation is the tried and tested way to treat the kidney cancer, it does have risks and complications, such as bleeding. The other two treatments are less intrusive to the patient, and are less complicated as they do not require such a large operation as having part of the kidney removed, but it is not known if they are as good at destroying all of the tumour, and whether or not patients who have their tumour destroyed with these new methods require further treatment in future.

In this study, the investigators are trying to determine if a large-scale study comparing these treatments is possible which is why this is called a feasibility study. The investigators are also looking at whether patients would be willing to be randomly assigned to a treatment group. The results of this study will then be compared to see how effective each of the treatments were and whether the number of patients who were happy to be randomly assigned to a treatment could be used to determine the number of patients required in a large-scale trial.

DETAILED DESCRIPTION:
This study will be a multicentre study to determine if it is possible to carry out a future trial comparing the effectiveness of two minimally invasive techniques to remove small kidney cancers, with the standard treatment of removing part of the diseased kidney. In this future study, participants will be randomly assigned (randomised) to one of these three treatment options. This current study will look at whether patients would be willing to be randomised to a treatment type, whether sufficient numbers for a larger trial would be likely to be recruited within a certain time period, and also to decide what aspects of the conduct and outcomes of each of the three treatment types would need to be recorded in a largescale trial to compare their effectiveness.

Eligible participants for this study will be identified and will be invited to take part in the study by their clinicians currently involved in their kidney cancer assessment. They would then receive information about the surgery treatment (removing the diseases part of the kidney) and one of the alternative treatment methods (destroying the kidney cancer tumour using either heat or by freezing) in the participating hospital. If the patient was interested in participating in the study, they will be asked to consent to be randomised to one of the two treatment types they were given the information about.

If a patient declines to be randomised to a treatment, they will be asked to participate in a series of interviews, to establish the reasons behind why they declined, such as if they had a preference for one of the treatments.

Those patients that consent to being randomised to one of the treatment arms will undergo a screening visit to confirm their eligibility for this study, and at this visit they will have a blood sampke taken and be asked to complete some questionnaires about their general health and how they feel. This is so that any questionnaires completed at a later date after treatment will be compared to how the patient responded before treatment, in order to look for any changes or improvements to the patients. Once they have been confirmed as eligible, they will be randomised to a treatment arm,, and a hospital appointment for their treatment will also be made at this time.

At the treatment visit, each patient will be admitted to hospital for their treatment as scheduled, and will be kept in hospital for the recommended duration after their operation. Those having the diseased part of the kidney removed will be kept in hospital for 35 days, those having their kidney cancer frozen using cryoablation will be kept in hospital for 2 days, and those having their kidney cancers destroyed using heat (radiofrequency ablation) will be kept in for one day.

As per standard care, this duration of time in hospital could vary if the patient experiences any unexpected complications. They will also have some blood samples taken at this visit to assess their kidney function.

All treatments will be given by a qualified specialist surgeon with extensive experience in the treatment they are giving the patient.

Three months after their treatment, each patient will be asked to return to their hospital for a followup visit. At this visit, the patients will be asked to complete the same questionnaires as was completed previously, as well as to undertake a CT scan to assess if the treatment they were given was successful and to determine if all the kidney cancer was removed or destroyed. This CT scan is for patients who undergo cryoablaton treatment only. Patients who undergo radiofrequency ablation treatment will have a CT scan one month after treatment. All patients will also have a blood sample taken at this visit to assess their kidney funtion.

Six months after their treatment, each patient will be asked to return to their hospital for a followup visit, at which point patients undergoing cryoablation treatment will once again have a CT scan to assess if their treatment remains a success, and to determine if all the kidney cancer is still destroyed or whether some of it has returned. They will be asked to complete the questionnaires from previous visits one more time, so as to compare how they feel and how their general health has improved or changed from previously.

Patients who undergo radiofrequency ablation treatment or cryoablation treatment will be required to attend for a further final visit within 2 weeks of their 6 month followup visit in order to have a kidney biopsy taken to determine if their treatment remains a success and all of the cancer mass has been destroyed.

After these six months, and five visit, the patient will return to their normal standard clinical followup visits, which they would be having whether they were on the study or not.

As well as these mentioned visits, some patients who consent to be randomised, will also be asked to consent to being involved in a series of interviews, at which times they will be asked general questions on how they feel in general and about the treatments they have received.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* ASA physical status classification system of 1 or 2
* Radiological confirmation of (>20 Hounsfield Unit) enhancing renal mass (< 4cm) or biopsy proven renal cancer
* CT abdomen/chest/pelvis with no enlarged nodes or distant metastases
* Patient has provided written informed consent for participation in the study prior to any study specific procedures

Exclusion Criteria:

* Coagulopathy
* Concomitant disease that would render the patient unsuitable for the study
* Presence of urosepsis
* Cancer which is completely buried in the kidney
* More than one small renal cancer mass
* Previous participation in this study
* Inability to give informed consent; carer/proxy assent will not be allowed in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who agree to trial registration and accept randomisation | 18 months
  To estimate the proportion of patients with renal masses < 4cm who agree to trial registration and accept randomisation to either partial nephrectomy or one of the ablative techniques

SECONDARY OUTCOMES:
SF-36 quality of life questionnaire | at 7 days of randomisation and at 3 to 6 months follow up
  To review responses and patients willingness to complete this questionnaire over the course of their involvement in the study
EQ-5D quality of life questionnaire | Within 7 days of randomisation, and at 3 and 6 months follow up
  To review responses and patient's willingess to complete this questionnaire during the course of their involvement in the study
FACT-G quality of life questionnaire | Within 7 days, and 3 and 6 month follow-up
  To review response and patients willingness to complete this questionnaire during the course of their involvement in the study
Hospital anxiety and depression questionnaire | Within 7 days, and 3 and 6 month follow up
  To review response and patients willingness to complete this questionnaire during the course of their involvement in the study
Differences in results in pre and post treatment CT scans | at 1, 3 and 6 months after surgery
  The timing of these CT scans is dependent on the treatment arm the patient is randomised to.
Effectiveness of treatment by a renal biopsy assessment | 6 months post treatment
  This renal biopsy is only applicable to patients undergoing ablative treatment
Response within qualitative interviews for patients who decline randomisation | Two to six weeks after recruitment interaction
Response within qualitative interviews following treatment | Eight to sixteen weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Soomro, Principal Investigator — Newcastle upon Tyne Hospitals NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - South Mead Hospital, Bristol
  - Gartnavel Hospital, Glasgow
  - Guys and St Thomas Hospital, London
  - St George's Hospital, London
  - Freeman Hospital, Newcastle upon Tyne